CLINICAL TRIAL: NCT02536261
Title: Dopamine Agonists Withdrawal Study of Invasive Prolactinomas Involving the Cavernous Sinus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhebao Wu (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other); First Hospital of China Medical University (Other); Beijing Tiantan Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Peking Union Medical College Hospital (Other); Huashan Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhebao Wu, Chief Physician, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Other Study IDs: WSIP-1586
Record Dates: First submitted 2015-08-15; First posted 2015-08-31 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Invasive Prolactinomas Involving the Cavernous Sinus
Keywords: Prolactinoma; dopamine agonist; withdrawal; cavernous sinus
MeSH Terms: conditions — Prolactinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood; urine; tumor specimens (if possible)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Withdrawal group: Withdrawal observation after reaching the withdrawal standard
- Continue treatment group: Continue treatment obsevation after reaching the withdrawal standard

SUMMARY:
The purpose of this study is to observe whether dopamine agonists can be safely withdrawn after the tumor volume and prolactin level of invasive prolactinomas involving the cavernous sinus have been effectively controlled through pharmacological treatment.

DETAILED DESCRIPTION:
For giant or large invasive prolactinomas involving the cavernous sinus, whether the drug can be safely withdrawn after the tumor volume and prolactin(PRL) level have been effectively controlled through pharmacological treatment still remains unknown. The study objects are patients with invasive prolactinomas involving the cavernous sinus, which were invaded the cavernous sinus to an extent corresponding to Grade III or IV, according to the classification scheme of Knosp and colleagues, who had undergone pharmacological treatment including bromocriptine or cabergoline. Observation will be started after drug withdrawal criteria are reached (PRL remains normal level for no less than two years; tumor volume has shrank more than 50%, and the distance is more than 5mm between tumor and optical nerve),the patients are randomized to withdrawal group or continue treatment group.Observational items include changes of PRL level, tumor volume as well as vision acuity and visual fields. If elevated PRL or tumor relapse is observed, pharmacological treatment will be restarted.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 15 and 70 years old, either sex;
2. Karnofsky performance status ≥ 70;
3. Patients who were suffered Invasive prolactinomas involving the cavernous sinus , referring to ①Serum prolactin level>200ng/ml, or >4000mIU/L;②enhanced Magnetic Resonance images confirm tumor invasion into cavernous sinus, i.e. Knosp grade Ⅲ or Ⅳ, and were treated by dopamine agonists treatment;
4. PRL remains normal level for no less than two years;
5. Tumor volume has shrank more than 50%, and the distance is more than 5mm between tumor and optical nerve;
6. The patient has signed the informed consent.

Exclusion Criteria:

1. Patients concomitantly taking the psychotropic drugs or other drugs causing elevated PRL ;
2. Patients with parkinson disease and is taking dopaminergic agents;
3. Patients with prolactinoma who received Gamma knife treatment;
4. Patients who use any dopamine receptor agonists other than bromocriptine and cabergoline;
5. Patients taking the other prolactinomas simultaneously;
6. pregnant or lactating women, or women preparing pregnant;
7. Patients with poor compliance, who cannot implement the program strictly.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: invasive prolactinomas involving the cavernous sinus
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on PRL level | Up to 2 years
  Record the result of PRL on every 3 month follow-up visit

SECONDARY OUTCOMES:
Change from baseline on tumor volume measured by enhanced pituitary Magnetic Resonance Imaging（MRI） | Up to 2 years
  Record the tumor volume from enhanced pituitary MRI on every 3 month follow-up visits
Change from baseline of visual acuity | Up to 2 years
  Record the Visual acuity on every 3 month follow-up visit
Change from baseline on 5 point visual field scale | Up to 2 years
  Record the Visual field scale on every 3 month follow-up visit, 0 = normal, no vision loss; 1 = one quadrant vision loss; 2 = two quadrants of vision loss; 3 = three quadrants of vision loss; 4 = four quadrants of vision loss but retain a central tubular vision; 5 = blind

CONTACTS AND LOCATIONS:
Overall Officials: Zhebao Wu, Medical PhD, Study Chair — Ruijin Hospital
Locations (8):
- China (8):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital of Chongqing, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hosipital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
The individual patient Data would not be shared to the third facility, but the sponsor hasn't decided whether to share the individual patient date to the other related studies hold by himself in the future.

REFERENCES:
- [Background] Wu ZB, Yu CJ, Su ZP, Zhuge QC, Wu JS, Zheng WM. Bromocriptine treatment of invasive giant prolactinomas involving the cavernous sinus: results of a long-term follow up. J Neurosurg. 2006 Jan;104(1):54-61. doi: 10.3171/jns.2006.104.1.54. PMID 16509147
- [Background] Wu ZB, Su ZP, Wu JS, Zheng WM, Zhuge QC, Zhong M. Five years follow-up of invasive prolactinomas with special reference to the control of cavernous sinus invasion. Pituitary. 2008;11(1):63-70. doi: 10.1007/s11102-007-0072-4. PMID 17917811